CLINICAL TRIAL: NCT03452293
Title: SUPERa Stenting After SUBintimal Crossing of TASC C-D Femoro-popliteal Lesions in CLI Patients
Acronym: SUPERSUBII
Status: Completed | Type: Observational
Sponsor: EndoCore Lab s.r.l. (Other)
Collaborators: Fondazione Italiana Vascolare (Other)
Responsible Party: Sponsor
Other Study IDs: EndoCore01
Record Dates: First submitted 2018-02-14; First posted 2018-03-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: PAD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stent Peripheral System — Peripheral PTA with Supera Stent implantation

SUMMARY:
The study will evaluate the safety and efficacy of subintimal Supera stenting in complex de novo or re-occlusive CTO (TASC C-D) lesions in patients with CLI. This study will be performed based on a rigorous sample size calculation, which will allow us to have the statistical power to validate our conclusions and therefore establish the generalizability of this strategy.

DETAILED DESCRIPTION:
The present study is designed as a prospective, open label, observational study.

The study will collect information about the medical care patients receive during their planned procedure. No additional testing or procedures will be done.

Patients elected for endovascular revascularization with SuperSub strategy will be asked their written consent to the use of their personal data.

Revascularization will be performed as per standard procedure of the sites. After discharge all patients will attend clinic visits at 30 days (±14 days), 6 months (±30 days), 12 months (±30 days) and 24 months (±30 days). Angiographic follow-up will be performed only in symptomatic patients, as clinically indicated and with the aim for a new treatment.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Patients with CLI and TASC C-D Fem-Pop CTO's
* Age ≥18 years
* Patient has signed an approved consent form
* Patients without previous stenting of the Fem-Pop segment

Angiographic Inclusion Criteria:

* Patent and hemodynamically normal iliac and common femoral arteries.
* At least one patent and healthy tibial vessel runoff to the foot.
* Patient has documented TASC C or D Fem-Pop CTO's prior to the study procedure
* Rutherford Category 4, 5 or 6
* Subintimal crossing of the occluded Fem-Pop vessels
* Supera Stenting From healthy to healthy arterial segment.

Exclusion Criteria:

* Patient unwilling or unlikely to comply with Follow-Up schedule
* Endoluminal crossing of the CTO
* Inability to stent from "healthy to healthy" arterial segments.
* Inability to re-enter within the pre-specified Ideal Landing Zone (IDL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by lower extremities artery disease and referred for the endovascular treatment of de novo or re-stenotic lesions (no in stent restenosis) in the femoro-popliteal arteries.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Primary Patency Rate | 24 months
  Primary Patency is defined as freedom from clinically driven TLR (CD-TLR) defined as repeat percutaneous intervention or surgical bypass graft to treat an angiographic significant restenosis (>50%) at the level of the treated lesion ±10 mm (proximally and/or distally)

SECONDARY OUTCOMES:
Freedom from Restenosis | 12 months
  Freedom from restenosis (diameter stenosis > 50%, determined by peak systolic velocity ratio (PSVR) >2.4 by duplex ultrasonography)
Freedom from Restenosis | 24 months
  Freedom from restenosis (diameter stenosis > 50%, determined by peak systolic velocity ratio (PSVR) >2.4 by duplex ultrasonography)
Composite of All Major Adverse Events | 12 Months
  Incidence of the composite of all Major Adverse Events
Composite of All Major Adverse Events | 24 Months
  Incidence of the composite of all Major Adverse Events
Incidence of Major Adverse Events | 12 months
  Incidence of Major Adverse Events
Incidence of Major Adverse Events | 24 months
  Incidence of Major Adverse Events
Stent integrity assessment | 12 months
  Stent integrity assessment will be evaluated with two oblique opposite projection X-ray images
Stent integrity assessment | 24 months
  Stent integrity assessment will be evaluated with two oblique opposite projection X-ray images
Primary Sustained Clinical Improvement | 6,12 and 24 months vs baseline
  Clinical Improvement as assessed by Rutherford Class changes
Quality of Life (EQ-5D-5L Questionnaire) | 6 months
  Quality of Life improvement as assessed by EQ-5D-5L Questionnaire Parameters [Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression] Values [(1) No Problems, (2) Slight Problems, (3) Moderate Problems, (4) Severe Problems, (5) Unable to] Value [1 - Best score, Value 5 - Worse Score]
Quality of Life improvement (SF12 Questionnaire) | 6 months
  Quality of Life improvement as assessed by SF12 Questionnaire Parameters [Overall Health, Physical health, Role and Physical health, Role and Mental health, Mental health] Values for Overall Health [ 1-Excellent, 2- Very Good, 3-Good, 4-Acceptable, 5-Poor] Values for Role and Physical health [ 1-Very limiting, 2-Partially limiting, 3-Not limiting] Values for Physical health [ 1-yes, 2-no], [1- best score] , [2-worse score] Values for Role and Mental health [ 1-yes, 2-no], [1- best score] , [2-worse score] Values for Mental Health [ 1-Excellent, 2- Very Good, 3-Good, 4-Acceptable, 5-Poor]
Quality of Life (EQ-5D-5L Questionnaire) | 12 months
  Quality of Life improvement as assessed by EQ-5D-5L Questionnaire Parameters [Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression] Values [(1) No Problems, (2) Slight Problems, (3) Moderate Problems, (4) Severe Problems, (5) Unable to] Value 1 - Best score, Value 5 - Worse Score
Quality of Life improvement (SF12 Questionnaire) | 12 months
  Quality of Life improvement as assessed by SF12 Questionnaire Parameters [Overall Health, Physical health, Role and Physical health, Role and Mental health, Mental health] Values for Overall Health [ 1-Excellent, 2- Very Good, 3-Good, 4-Acceptable, 5-Poor] Values for Role and Physical health [ 1-Very limiting, 2-Partially limiting, 3-Not limiting] Values for Physical health [ 1-yes, 2-no], [1- best score] , [2-worse score] Values for Role and Mental health [ 1-yes, 2-no], [1- best score] , [2-worse score] Values for Mental Health [ 1-Excellent, 2- Very Good, 3-Good, 4-Acceptable, 5-Poor]
Quality of Life (EQ-5D-5L Questionnaire) | 24 months
  Quality of Life improvement as assessed by EQ-5D-5L Questionnaire Parameters [Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression] Values [(1) No Problems, (2) Slight Problems, (3) Moderate Problems, (4) Severe Problems, (5) Unable to] Value 1 - Best score, Value 5 - Worse Score
Quality of Life improvement | 24 months
  Quality of Life improvement as assessed by SF12 Questionnaire Parameters [Overall Health, Physical health, Role and Physical health, Role and Mental health, Mental health] Values for Overall Health [ 1-Excellent, 2- Very Good, 3-Good, 4-Acceptable, 5-Poor] Values for Role and Physical health [ 1-Very limiting, 2-Partially limiting, 3-Not limiting] Values for Physical health [ 1-yes, 2-no], [1- best score] , [2-worse score] Values for Role and Mental health [ 1-yes, 2-no], [1- best score] , [2-worse score] Values for Mental Health [ 1-Excellent, 2- Very Good, 3-Good, 4-Acceptable, 5-Poor]
Amputation Rates | 1 month
  Major and Minor amputations
Amputation Rates | 6 months
  Major and Minor amputations
Amputation Rates | 12 months
  Major and Minor amputations
Amputation Rates | 24 months
  Major and Minor amputations

OTHER OUTCOMES:
Cost-efficiency analysis | 12 months
  Cost-efficiency analysis based on the comparison of the yearly procedural related costs and hospital stay(s) between patients treated with the SUPERSUB strategy, vs a propensity-matched historical cohort of patients with the same type of lesions (TASC C-D), treated by PTA alone, after subintimal crossing.
Cost-efficiency analysis | 24 months
  Cost-efficiency analysis based on the comparison of the yearly procedural related costs and hospital stay(s) between patients treated with the SUPERSUB strategy, vs a propensity-matched historical cohort of patients with the same type of lesions (TASC C-D), treated by PTA alone, after subintimal crossing.
Technical success | 1 month
  Technical success defined as achievement of a final in-lesion residual diameter stenosis of ≤30% as determined by the angiographic core lab
Clinical success | 1 month
  Clinical success defined as technical success without the occurrence of major adverse events
Procedural success | 1 month
  Procedural success defined as lesion success without the occurrence of major adverse events
ABI index or transcutaneous oxymetry (TcPO2) improvement | 6 and 12 months vs baseline
  Improve in the ABI index or transcutaneous oxymetry (TcPO2)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Salomone, MD, Study Director — EndoCore Lab; Mariano L Palena, MD, Study Chair — Casa di Cura Abano Terme; Larry J Diaz, MD,PhD, Study Chair — Metro Health Hospital
Locations (15):
- Metro Health Hospital, Wyoming, Michigan, United States
- Instituto Medico CENICLAR, Unidad Sanatorio de la Mujer, Rosario, Santa Fe Province, Argentina
- Italy (12):
  - Ospedale di Avezzano, Avezzano, AQ
  - Clinica San Michele, Maddaloni, CE
  - A.O.U. Policlinico Vittorio Emanuele, Catania, CT
  - A.O. Cardinale Panico, Tricase, LE
  - Casa di Cura Abano Terme, Abano Terme, Padova
  - A.O.U. Santa Maria della Misericordia, Perugia, PG
  - Policlinico Tor Vergata, Roma, RM
  - A.O. San Giovanni Addolorata, Roma, RM
  - A.O.U. di Sassari, Sassari, SS
  - Ospedale San Antonio Abate, Erice, TP
  - Azienda Ospedaliera Santa Maria di Terni, Terni, TR
  - AORN Antonio Cardarelli, Napoli
- London North West HealthCare NHS Trust, London, England, United Kingdom